CLINICAL TRIAL: NCT03542357
Title: The Effect of Sumatriptan and Placebo on CGRP Induced Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Katrine Falkenberg, Medical doctor, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-16000065
Record Dates: First submitted 2017-10-20; First posted 2018-05-31 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Calcitonin Gene-Related Peptide; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sumatriptan (Active Comparator): headache is induced with CGRP. This headache is treated double-blinded with 1 tablet of sumatriptan 50 mg as a pre-treatment
  Interventions: Drug: Calcitonin Gene Related Peptide; Drug: Sumatriptan 50 mg
- Placebo (Placebo Comparator): headache is induced with CGRP. This headache is treated double-blinded with 1 tablet of placebo as a pre-treatment
  Interventions: Drug: Calcitonin Gene Related Peptide; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Calcitonin Gene Related Peptide — CGRP is given both study days to induce headache. One day the headache is treated with placebo and the other day with sumatriptan
  Other Names: CGRP
Drug: Sumatriptan 50 mg — CGRP is given both study days to induce headache. One day the headache is treated with placebo and the other day with sumatriptan
  Other Names: Imigran
  Arms: Sumatriptan
Drug: Placebo Oral Tablet — CGRPis given both study days to induce headache. One day the headache is treated with placebo and the other day with sumatriptan
  Arms: Placebo

SUMMARY:
To develop a pragmatic migraine model the investigators will induce headache in healthy volunteers and in patients with migraine without aura with aCalcitonine Gene Related Peptide (CGRP). If the headache responds to sumatriptan, the model can be used to test new drug candidates.

DETAILED DESCRIPTION:
There remains a great need for more effective anti-migraine drugs with fewer side effects. Human experimental models are valuable in early phase development of new anti-migraine drugs but useful models have not yet been developed. The investigators' group has shown that Calcitonine Gene Related Peptide (CGRP) induce headache/migraine in both healthy volunteers and in patients with migraine without aura (MO). To validate this model, the headache must respond to specific migraine treatment with sumatriptan.

Hypothesis: CGRP induces a migraine-like headache in both healthy subjects and in MO-patients and induced headache responds to a specific anti migraine drug; sumatriptan.

Aim: Developing a pragmatic and valid model for the testing of new anti-migraine drugs.

ELIGIBILITY:
Inclusion criteria:

Healthy:

Healthy subjects of both sexes Age 18-60 years Weight 45-95 kg. Females were requested to use effective contraception.

Migraine patients:

Migraine patients who meet IHS criteria for migraine with or without aura of both sexes 18-60 years 45-95 kg.

Exclusion Criteria:

Healthy:

Any type of headache (except episodic tension-type headache < 1 day per week) Serious somatic or psychiatric disease Pregnancy Intake of daily medication (except oral contraceptives).

Migraine patients:

Any other type of headache then migraine without aura (except episodic tension-type headache < 1 day per week) Serious somatic or psychiatric disease Pregnancy Intake of daily medication (except oral contraceptives) Triptan non-responders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
AUC after infusion | 1 year
  The investigators will assess the outcome measures 1 year after the beginning of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No